CLINICAL TRIAL: NCT01353222
Title: A Randomized, Phase 2, Open-label Study Evaluating DN24-02 as Adjuvant Therapy in Subjects With High Risk HER2+ Urothelial Carcinoma
Brief Title: DN24-02 as Adjuvant Therapy in Subjects With High Risk HER2+ Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N10-1
Record Dates: First submitted 2011-05-04; First posted 2011-05-13 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Urothelial Carcinoma
Keywords: Bladder cancer; Renal pelvis cancer; Ureteral cancer; Urethral cancer; Bladder; Renal pelvis; Ureter; Urethra; Immune therapy; Immunotherapy; Vaccine; Dendritic cells; Antigen-presenting cells; Antigen presenting cells; Cancer vaccine; Urothelial carcinoma; Urothelial neoplasms; Neoplasms by site; Neoplasms
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms; Neoplasms by Site; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DN24-02 (Experimental): Subjects received infusion of DN24-02, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: DN24-02
- Standard of Care (Other): Subjects randomized to the control arm were treated per standard of care, which in this patient population is generally observation, as there is currently no evidence that treatment with non-cisplatin containing chemotherapy is beneficial in the adjuvant setting for this patient population.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: DN24-02 — DN24-02 is an autologous cellular immunotherapy product designed to stimulate an immune response against HER2/neu. It consists of autologous peripheral blood mononuclear cells (PBMCs), including antigen presenting cells (APCs), which are activated ex vivo with a recombinant fusion protein, BA7072.
  Arms: DN24-02
Other: Standard of Care — Observation only until documentation of disease recurrence.
  Arms: Standard of Care

SUMMARY:
This study was conducted to examine survival, disease-free survival, safety, and the magnitude of the immune response induced following administration of DN24-02 in subjects with HER2+ urothelial carcinoma.

DETAILED DESCRIPTION:
Multicenter, open-label, Phase 2 study. Subjects were randomized to either the investigational product, DN24-02, or to standard of care. Subjects randomized to the experimental arm received DN24-02 at 2-week intervals, for a total of 3 infusions. The study evaluated survival, disease-free survival, safety and the magnitude of the immune response between these 2 subject groups.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic evidence of urothelial carcinoma, based on local pathology report.
* High risk urothelial carcinoma, in subjects with or without prior neoadjuvant chemotherapy, defined as positive lymph node status (N+), or pathological stage ≥ pathological tumor (pT2) in patients who either have negative lymph node status (N0) or have no evaluable lymph nodes (Nx).
* Radical surgical resection was performed ≤ 84 days (12 weeks) prior to registration.
* No evidence of residual disease or metastasis following surgical resection which includes: absence of invasive cancer at the margins in the surgical specimens and confirmation by CT scan of chest, abdomen and pelvis obtained at least 28 days following surgical resection and ≤ 28 days prior to registration.
* HER2/neu tissue expression ≥ 1+ by immunohistochemistry (IHC). Available biopsy specimens from the primary tumor and involved lymph nodes are be submitted to the central pathology laboratory prior to registration for confirmation of HER2/neu tissue expression.
* Last neoadjuvant chemotherapy treatment administered at least 60 days prior to registration.
* Left ventricular ejection fraction ≥ 50% on multigated acquisition (MUGA) scan or echocardiogram obtained at least 28 days following surgery and ≤ 28 days prior to registration.
* Women of child-bearing potential have a negative serum pregnancy test result ≤ 28 days prior to registration and agree not to breastfeed during investigational treatment with DN24-02 and for 28 days following the final infusion of DN24-02.
* All males and premenopausal females who have not been surgically sterilized have agreed to practice a method of birth control considered by the Investigator to be effective and medically acceptable for at least 14 days prior to registration, throughout treatment, and for 28 days following the final infusion of DN24-02.
* Adequate hematologic, renal, and liver function.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* A history of stage III or greater non-urothelial cancer. Exceptions include: Subject with basal or squamous cell skin cancers that has been adequately treated who are disease-free at the time of registration. Subjects who have been disease-free and off treatment for ≥ 10 years at the time of registration.
* A history of stage I or II non-urothelial cancer. Exceptions include: Subjects who have been disease-free and off treatment for ≥ 3 years at the time of registration. Subjects with incidental prostate cancer diagnosed at the time of cystoprostatectomy. Subjects with basal or squamous cell skin cancer.
* Partial cystectomy in the setting of bladder cancer primary tumor.
* Partial nephrectomy in the setting of renal pelvis primary tumor.
* Adjuvant systemic therapy for urothelial or prostatic carcinoma following surgical resection.
* Adjuvant radiation therapy for urothelial or prostatic carcinoma following surgical resection.
* Incidental prostate cancer with detectable post-operative (radical cystoprostatectomy) prostate specific antigen (PSA) levels ≤ 28 days prior to registration.
* Any major surgery (e.g., surgery requiring general anesthesia) ≤ 28 days prior to registration.
* Systemic treatment on any investigational clinical trial ≤ 28 days prior to registration.
* Systemic glucocorticoid or immunosuppressive therapy use ≤ 28 days prior to registration.
* Any infection requiring parenteral antibiotic therapy or causing fever (i.e., temperature > 100.5°F or > 38.1°C) ≤ 7 days prior to registration.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to DN24-02 or Granulocyte-macrophage colony-stimulating factor (GM-CSF).
* Any medical intervention, has any other condition, or has any other circumstance which, in the opinion of the Investigator or the Dendreon Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (60):
- United States (60):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Genesis Research, San Diego, California
  - Stanford University Hospital, Stanford, California
  - University of Colorado, Anschutz Cancer Pavilion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Neag Comprehensive Cancer Center/University of Connecticut Health Center, Farmington, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Urological Research Network, Hialeah, Florida
  - University of Miami Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Emory Department of Urology, The Emory Clinic Inc, Emory University Hospital, Atlanta, Georgia
  - American Red Cross, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Kansas City Urology Care, Overland Park, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Michigan Institute of Urology, Troy, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - GU Research Center, LLC, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Clinical Cancer Center, NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Mount Sinai School of Medicine Department of Urology, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Associated Medical Professionals of NY, PLLC, Oneida, New York
  - University of Rochester Medical Center, Rochester, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - UNC Health Care, NC Cancer Hospital, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - TriState Urologic Services PSC, Inc. dba TUG Research, Cincinnati, Ohio
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Jewish Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, James Cancer Hospital, Martha Morehouse Medical Plaza, Ohio State University Dept of Urology, Columbus, Ohio
  - Urologic Specialists of Oklahoma, Tulsa, Oklahoma
  - OHSU Knight Cancer Institute Hematology Oncology, Beaverton, Oregon
  - Providence Medical Center, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Urology Health Specialists, LLC, Bryn Mawr, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - UW Medical Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Subjects randomized to the control arm were treated per standard of care, which in this patient population is generally observation, as there is currently no evidence that treatment with non-cisplatin-containing chemotherapy is beneficial in the adjuvant setting for this patient population.
Period: Overall Study
Arm/Group | DN24-02 | Standard of Care
Started | 70 | 72
DN24-02 Arm ≥1 Leukapheresis (Safety population for the DN24-02 arm.) | 67 | 0
Standard Care Arm ≥1 Post-baseline Visit (Safety population for the Standard of Care arm.) | 0 | 72
Completed | 0 | 0
Not Completed | 70 | 72
Not completed — Death | 30 | 30
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Study Terminated | 31 | 37
Not completed — Site closed research department | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | DN24-02 | Standard of Care | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (10.81) | 66.4 (10.09) | 66.0 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 52 | 53 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 65 | 70 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 72 | 142
Body weight [Mean (Standard Deviation); unit: kilograms] — Population: Baseline weight for one subject in standard of care group is missing.
  kilograms
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 80.770 (18.3080) | 82.115 (17.9330) | 81.448 (18.0679)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead Population: Baseline ECOG data is missing for one subject in each group.
  Participants
    ECOG 0=Fully Active; No restrictions: number analyzed (Participants) | 69 | 71 | 140
    ECOG 0=Fully Active; No restrictions | 42 | 38 | 80
    ECOG 1= Restricted Strenuous Activity: number analyzed (Participants) | 69 | 71 | 140
    ECOG 1= Restricted Strenuous Activity | 24 | 31 | 55
    ECOG 2=Ambulatory, capable of self-care; no work: number analyzed (Participants) | 69 | 71 | 140
    ECOG 2=Ambulatory, capable of self-care; no work | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death due to any cause.
  *This study was terminated early due to administrative reasons.
Time Frame: Subjects will be followed from baseline through the remainder of their lives or until study completion (approximately 60 months)
Population: Intent to Treat (ITT) population.
  *This study was terminated early due to administrative reasons.
Measure: Median (Full Range); unit: Months
Groups:
- Standard of Care: Subjects randomized to the control arm were treated per standard of care, which in this patient population is generally observation, as there is currently no evidence that treatment with non-cisplatin containing chemotherapy is beneficial in the adjuvant setting for this patient population.
  Standard of Care: Standard of care
Arm/Group | DN24-02 | Standard of Care
Number analyzed (Participants) | 70 | 72
Months | 17.2 [0.1 to 42.4] | 18 [0.3 to 40.2]
Statistical Analysis 1: Comparison: DN24-02 vs Standard of Care; Test type: Superiority; p = 0.6188, From a stratified log-rank test, stratif; Hazard Ratio (HR) = 1.141, 95% CI 2-sided [0.679 to 1.918] — Cox regression model with treatment as the independent variable, stratified by randomization strata. Hazard ratio with control as reference

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of registration through investigator-assessed disease recurrence or 30 days following the final infusion of DN24-02, whichever occurred later.
Description: Adverse events are reported in the safety population. The safety population was defined as all subjects in the treatment arm who underwent at least 1 leukapheresis and all randomized control subjects with at least 1 post-baseline safety assessment or visit.
Arm/Group | DN24-02 | Standard of Care
All-Cause Mortality (participants affected / at risk) | 30/67 | 30/72
Serious Adverse Events (participants affected / at risk) | 20/67 | 17/72
Other Adverse Events (participants affected / at risk) | 64/67 | 52/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DN24-02 (N=67) | Standard of Care (N=72)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 4 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MEDICAL OBSERVATION (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
FOLLICLE CENTRE LYMPHOMA, FOLLICULAR GRADE I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 (3) | 1 (1)
URETERIC STENOSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLADDER IRRIGATION (Surgical and medical procedures) | 1 (1) | 0 (0)
BLADDER REPAIR (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
SHOULDER OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
ANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DN24-02 (N=67) | Standard of Care (N=72)
ANAEMIA (Blood and lymphatic system disorders) | 8 (8) | 5 (6)
CONSTIPATION (Gastrointestinal disorders) | 14 (15) | 10 (10)
NAUSEA (Gastrointestinal disorders) | 18 (27) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (9) | 9 (9)
VOMITING (Gastrointestinal disorders) | 10 (17) | 7 (7)
DIARRHOEA (Gastrointestinal disorders) | 12 (13) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 4 (4)
FATIGUE (General disorders) | 26 (36) | 15 (17)
CHILLS (General disorders) | 24 (37) | 1 (1)
PYREXIA (General disorders) | 17 (20) | 5 (10)
OEDEMA PERIPHERAL (General disorders) | 7 (9) | 3 (5)
PAIN (General disorders) | 7 (10) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 4 (6) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 9 (25)
NASOPHARYNGITIS (Infections and infestations) | 7 (7) | 5 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 2 (2)
WEIGHT DECREASED (Investigations) | 6 (6) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 (15) | 6 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (9) | 10 (14)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (8)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
HEADACHE (Nervous system disorders) | 13 (16) | 4 (4)
DIZZINESS (Nervous system disorders) | 5 (6) | 4 (4)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 (8) | 1 (2)
INSOMNIA (Psychiatric disorders) | 4 (4) | 4 (4)
HAEMATURIA (Renal and urinary disorders) | 7 (8) | 6 (6)
INCONTINENCE (Renal and urinary disorders) | 2 (2) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5)
RASH (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
HYPOTENSION (Vascular disorders) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentation relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.